CLINICAL TRIAL: NCT04628975
Title: Evaluation of the Efficacy of Transillumination on Peripheral Venous Line Placement in Patients With a Difficult Vascular Approach Who Are Managed in the Emergency Department.
Brief Title: PeRfusion Emergency VEiNlite Transillumination
Acronym: PREVENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00891-38
Record Dates: First submitted 2020-10-21; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-08

CONDITIONS: Emergencies; Toxicomania; Hypotension; Obesity; Cachexia; Hypothermia
Keywords: adult; peripheral venous approach; emergency; transillumation
MeSH Terms: conditions — Emergencies; Hypotension; Obesity; Cachexia; Hypothermia

STUDY DESIGN:
Intervention Model Description: multi-center prospective randomized cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with transillumination (Experimental): The nurses will use the Transillumination method for a period P1. Then these same nurses will use the control method (without transillumination) for a period P2.
  Interventions: Device: transillumination dispositif
- without transillumination (control method) (No Intervention): The nurses will use the control method for a period P1. Then these same nurses will use the Transillumination method for a period P2.

INTERVENTIONS:
Device: transillumination dispositif — infrared light
  Arms: with transillumination

SUMMARY:
When taking care of an emergency patient (Emergency Reception Service: UAS and Urgent Medical Assistance Service: SAMU), the installation of a peripheral venous route (VVP) is an important step. The benchmark method is the most widely used technique. This vascular access will allow the necessary therapy to be delivered quickly and efficiently. This can be difficult and sometimes doomed to failure for reasons related both to the patient (venous capital not very visible / felt or limited due to the profile of the patient), or sometimes also for reasons related to the patient. environment (limited lighting, difficult patient access). The only current alternatives lie in the use of a device such as the Intra-Bone Device (IID) or the installation of a central venous line. On the other hand, these alternatives are particularly invasive and / or very algogenic.

There are other techniques, which are more affordable and "transportable" outside the hospital. Indeed, trans-illumination with a very short training seems to be a particularly interesting alternative. It allows, thanks to LEDs in contact with the skin, to backlight the superficial veins.

It is proposed through this project to evaluate this tool for a category of patients considered "difficult" to infuse, both within hospital and outside hospital.

The main objective of the study is to assess the effectiveness of the transillumination device, compared to the absence of such a device, on the placement of a peripheral venous line (PVP) in patients with a difficult vascular approach and managed in the emergency room and whose clinical condition does not require the installation of an intraosseous device.

This is a multicenter, prospective, controlled, randomized and open clinical study, according to a cross-over design. The intervention evaluated is the placement of a PVR using the trans-illumination device. The control intervention is the placement of a PVR without this device, according to the reference method, which is the benchmark method.

400 patients presenting to the emergency room will be included in the centers of Nancy, Toul and Pont-à-Mousson.

Depending on their randomization group, nurses will perform peripheral venous insertion by the transillumination method or by the control method.

ELIGIBILITY:
Inclusion Criteria:

>= 18 years old

* extrem body mass index
* hypotension
* toxicomania
* limited ponction site
* hypotherm patient
* dehydrated patient
* generalized edema
* non-supportive environment

Exclusion Criteria:

* parturient / pregnant female / breastfeeding mother
* unemancipated minor
* adults under legal protection
* person under judicial protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients for whom peripheral venous vein placement was successful on the first attempt | immediately after procedure

SECONDARY OUTCOMES:
number of attempts before successful venous line placement | during the procedure
patient pain | during the procedure
  The patient's pain is measured by the digital pain scale (scale ranging from 0 (no pain) to 10 (intolerable pain)).
nurse stress | during the procedure
  Nurse stress is measured by the digital stress scale (scale ranging from 0 (no stress) to 10 (intolerable stress)).
The caliber of the peripheral venous route | during the procedure
  measured by the type of catheter gauge used

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Staszewski, Principal Investigator — CH Pont à Mousson